CLINICAL TRIAL: NCT04292873
Title: Investigating the Effects of Enteral Supplement of Vitamin D in Critically Ill Patients With Vitamin D Deficiency
Brief Title: Effects of Enteral Supplement Vitamin D Incritically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201902073MIPA
Record Dates: First submitted 2020-03-01; First posted 2020-03-03 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Vitamin D Deficiency; Critical Illness
Keywords: Vitamin D Deficiency, critical Illness
MeSH Terms: conditions — Vitamin D Deficiency; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Vitamin D (Experimental): Enteral supplement of 569,600 IU vitamin D
  Interventions: Other: Vitamin D supplement

INTERVENTIONS:
Other: Vitamin D supplement — Enteral supplement of 569,600 IU vitamin D
  Arms: Vitamin D

SUMMARY:
At present, there is no clinical reference data on how much the concentration of calcifediol in the blood increases after supplementing with vitamin D for Taiwanese ICU patients. This study aims to investigate the effects of enteral supplementation of vitamin D in critically ill patients with vitamin D deficiency. The results of the study are expected to provide clinical reference data to intensivists to select adequate dosage of vitamin D supplementation for their patients with vitamin D deficiency.

This is a multi-center, randomized clinical trial. ICU patients will receive vitamin D level examination. If the subject's blood calcifediol concentration is less than 20 ng / mL, the subject will be included in this clinical trial. Patients who are suitable to enteral supplement of vitamin D will be randomly divided to group Control (no vitamin D supplement) and group Vitamin D (enteral supplement of 569,600 IU vitamin D). The vitamin D level will be measures at specific time points.

DETAILED DESCRIPTION:
Vitamin D deficiency patients have longer hospital stays, higher medical expenditures, and higher sepsis-related mortality. The preliminary results of 145 ICU patients of the Northern Medical Centers in Taiwan in our ongoing multicenter clinical trial showed that the mean calcifediol concentration was about 20.9 ng/mL, much lower than the normal value of 30-60 ng/ml. An Austrian randomized clinical trial has shown that supplementation of high-dose vitamin D in critically ill patients with vitamin D deficiency can reduce patient mortality, so it is important to treat critically ill patients with vitamin D deficiency. At present, there is no clinical reference data on how much the concentration of calcifediol in the blood increases after supplementing with vitamin D for Taiwanese ICU patients. This study aims to investigate the effects of enteral supplementation of vitamin D in critically ill patients with vitamin D deficiency. The results of the study are expected to provide clinical reference data to intensivists to select adequate dosage of vitamin D supplementation for their patients with vitamin D deficiency.

This is a multi-center, randomized clinical trial. ICU patients will receive vitamin D level examination. If the subject's blood calcifediol concentration is less than 20 ng / mL, the subject will be included in this clinical trial. Patients who are suitable to enteral supplement of vitamin D will be randomly divided to group Control (no vitamin D supplement) and group Vitamin D (enteral supplement of 569,600 IU vitamin D). The vitamin D level will be measures at specific time points. The patients' diagnosis, vital signs, laboratory data, 30-day survival, and 90-day survival will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients in intensive care units
* blood calcifediol concentration less than 20 ng / mL
* suitable for enteral feeding
* no ileus, vomit, or diarrhea

Exclusion Criteria:

* younger than 20 years old
* receive high dose vitamin D within 4 weeks (> 3000 IU pre day)
* hypercalemia ( > 2.6 mmol/L)
* body weight < 45 or > 90 kg
* admitted to intensive care unit before this admission within 3 months
* have diseases as follows: parathyroid disease, rickets, or liver cirrhosis - Child C
* diagnosed with renal stone, tuberculosis, or sarcoidosis
* Non-native speaker

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Vitmain D level | 7 days
  blood level of vitamin D

SECONDARY OUTCOMES:
Vitmain D level | 14 days
  blood level of vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang AY, Yeh YC, Cheng KH, Han YY, Chiu CT, Chang CC, Wang IT, Chao A. Efficacy and safety of enteral supplementation with high-dose vitamin D in critically ill patients with vitamin D deficiency. J Formos Med Assoc. 2025 Apr;124(4):355-360. doi: 10.1016/j.jfma.2024.05.005. Epub 2024 May 10. PMID 38729818